CLINICAL TRIAL: NCT02196740
Title: Randomized Controlled Research of the Application of Triple Antibiotic Paste in Primary Teeth With
Brief Title: Research of the Application of Triple Antibiotic Paste in Primary Teeth With Pericpical Periodontitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Lin Jiacheng (Other)
Responsible Party: Sponsor-Investigator, Lin Jiacheng, Research Associate, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Tri-antibiotic-2014
Record Dates: First submitted 2014-07-17; First posted 2014-07-22 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Periapical Diseases
Keywords: periapical periodontitis,primary teeth
MeSH Terms: conditions — Periapical Diseases; Periapical Periodontitis | interventions — Creosote

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- creosote (Active Comparator): Creosote ，once，three weeks Triple Antibiotic Paste ，none
  Interventions: Drug: creosote
- Triple Antibiotic Paste (Experimental): Triple Antibiotic Paste,once,three weeks creosote,none
  Interventions: Drug: Metronidazole-Ciprofloxacin gatifloxacin-Clindamycin paste

INTERVENTIONS:
Drug: Metronidazole-Ciprofloxacin gatifloxacin-Clindamycin paste — Pulp removal,Root canal irrigation and disinfection,
  Arms: Triple Antibiotic Paste
Drug: creosote — Pulp removal,Root canal irrigation and disinfection
  Other Names: oily liquid obtained by distillation of wood tar
  Arms: creosote

SUMMARY:
The triple antibiotic paste is widely used in young permanent teeth and permanent teeth root canal therapy with excellent antiantimicrobial effect.We hypothesize that its application in the treatment of periapical periodontitis of deciduous teeth is superior to other drugs currently in use as creosote.

DETAILED DESCRIPTION:
We design to collect a group of patients presenting primary teeth with periapical periodontitis in certain criterion. We will divide the patients into two groups randomly.One group will get treated with triple antibiotic paste while the other with creosote.We want to evaluate the short-term and long-term effects of the two groups to get a conclusion of the clinical value of triple antibiotic paste.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of periapical periodontitis
* must be primary teeth
* must be 3~8 years old
* the permanent tooth germ is complete and didnot be involved

Exclusion Criteria:

* blood disease
* residual root that is advised to extract
* serious periodontitis
* allergy to the triple antibiotic paste

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2013-06; Primary Completion 2014-12 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Evidence of lesion healing confirmed by cone beam computed tomography and X-rays | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jiacheng Lin, Study Chair — Guanghua hospital of stomotology,Sun Yat-sen University
Locations (1):
- Jicheng Lin, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Bezgin T, Yilmaz AD, Celik BN, Sonmez H. Concentrated platelet-rich plasma used in root canal revascularization: 2 case reports. Int Endod J. 2014 Jan;47(1):41-9. doi: 10.1111/iej.12144. Epub 2013 Jun 17. PMID 23772873
- [Background] Nagata JY, Gomes BP, Rocha Lima TF, Murakami LS, de Faria DE, Campos GR, de Souza-Filho FJ, Soares Ade J. Traumatized immature teeth treated with 2 protocols of pulp revascularization. J Endod. 2014 May;40(5):606-12. doi: 10.1016/j.joen.2014.01.032. Epub 2014 Mar 6. PMID 24767551
- [Background] Nagata JY, Soares AJ, Souza-Filho FJ, Zaia AA, Ferraz CC, Almeida JF, Gomes BP. Microbial evaluation of traumatized teeth treated with triple antibiotic paste or calcium hydroxide with 2% chlorhexidine gel in pulp revascularization. J Endod. 2014 Jun;40(6):778-83. doi: 10.1016/j.joen.2014.01.038. Epub 2014 Apr 29. PMID 24862703